CLINICAL TRIAL: NCT07154576
Title: Central Sensitization Inventory and Symptoms of Pelvic Floor Dysfunctions
Status: Not yet recruiting | Type: Observational
Sponsor: Żelazna Medical Centre, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: PN/99/2024
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Floor Dysfunctions
Keywords: pelvic floor dysfunctions; pelvic organ prolapse; central sensitization inventory
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- women attending gynecology outpatient clinic

SUMMARY:
The goal of this observational study is to assess the values of Central Sensitization Inventory in women in a gynecology outpatient clinic. The main question it aims to answer is:

Is there a relationship between outcomes of Central Sensitization Inventory and symptoms of pelvic floor dysfunctions reported by the patients?

Participants will complete questionnaires: Central Sensitization Inventory and questionnaires assessing pelvic floor dysfunctions and their impact on quality of life (PFDI-20, PFIQ-7, PISQ-12).

DETAILED DESCRIPTION:
Background: Pelvic floor dysfunctions are common disorders negatively impacting women's quality of life. However, there are differences when assessing prevalence due to the type of assessment. Prevalence of pelvic organ prolapse ranges between 1-65% of women; when assessing prevalence depending on symptoms, it can be 1-31%, but using anatomical examination, 1-50%, and finally, both of them - 20-65%.

Factors that are responsible for these discrepancies are still unknown. There are suggestions about correlations between central sensitivity syndrome (CSS) and differences in symptoms reported by patients, and the effect of surgical treatment.

Objectives: The aim of this study is to assess the values of Central Sensitization Inventory in women in gynecology outpatient clinic. Moreover, to examine if there is a relationship between those outcomes and symptoms of pelvic floor dysfunctions reported by the patients.

Material and methods: Women attending gynecological outpatient clinics will be invited to this study. Participants will be asked to complete the following questionnaires: Central Sensitization Inventory (CSI) and questionnaires assessing pelvic floor dysfunctions and their impact on quality of life (PFDI-20, PFIQ-7, PISQ-12). Pelvic organ prolapse will be assessed using the POP-Q scale.

Expected results: To our knowledge, this will be the first study of this type conducted in Poland. Obtained results will provide preliminary, descriptive information on values of the Central Sensitization Inventory and questionnaires assessing pelvic floor dysfunctions and their impact on quality of life. Data from this study may become a starting point for further, larger projects aimed at improving treatment of pelvic floor dysfunctions, including both physiotherapy and surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* women attending gynecological outpatient clinics
* Agreement to participate
* Good command of spoken and written Polish

Exclusion Criteria:

* age below 18
* women who have undergone surgical treatment of pelvic organ prolapse or urinary incontinence
* Lack of consent to participate in the study
* Lack of good command of spoken and written Polish
* pregnancy
* women up to 6 months postpartum

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women attending gynecology outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 359 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Central Sensitization Inventory (CSI) | baseline measurement
  questionnaire which is divided into two parts A and B. The first contains 25 questions about symptoms, and 5 answers scored 0-4 for each, allowing for a score from 0 to 100. Part B contains information about the occurrence of diseases in the past
Polish version of the Pelvic Floor Distress Inventory (PFDI-20) | baseline measurement
  Condition-specific questionnaire that will be used to assess how pelvic floor disorders affect quality of life. It consists of 3 scales, 20 questions. Every scale is scored from 0- no distress to 100 - the greatest distress. The scores from the 3 scales are summarized to achieve summary score (0-300)
Pelvic Organ Prolapse Quantification (POP-Q) system | baseline measurement
  It is an objective, site-specific system that allows one to describe, quantify and stage pelvic support in women on a scale 0-4, 0 indicates no prolapse, while 4 indicates the most severe stage of pelvic organ prolapse.
Polish version of the Pelvic Floor Impact Questionnaire short form 7 (PFIQ-7) | baseline measurement
  Condition-specific questionnaire that will be used to assess the impact of pelvic floor disorders on quality of life (daily activities, relationships and emotions). It consists of 3 scales which are scored 0-100. The results from the 3 scales are summarized to achieve the summary score (0-300). Higher numbers indicate greater impact.
Polish version of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) | baseline measurement
  A condition-specific tool to assess sexual function in women with pelvic floor disorders. It contains 12 questions, where responses are graded on a five-point Likert scale ranging from 0 (always) to 4 (never). 48 is the maximum score, where higher scores indicate better sexual function.

CONTACTS AND LOCATIONS:
Locations (1):
- Żelazna Medical Center, Warsaw, Poland